CLINICAL TRIAL: NCT02371200
Title: A Pivotal, Phase III Trial of Detecting Generalized Tonic-Clonic Seizures With a Seizure Detection and Warning System (System Version 1.5) in Epilepsy Patients
Brief Title: Detecting Generalized Tonic-Clonic Seizures With a Seizure Detection and Warning System in Epilepsy Patients
Status: Completed | Type: Observational
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Other Study IDs: GTC-1.5-09.2015
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy; Generalized Tonic-Clonic Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Sentinel Seizure Detection and Warning System: This study will compare accuracy of seizure detection by the study device to simultaneously collected data of seizure detection by video EEG.
  Interventions: Device: Brain Sentinel Seizure Detection and Warning System

INTERVENTIONS:
Device: Brain Sentinel Seizure Detection and Warning System — The detection device is worn on the bicep brachii muscles and is intended to alert a remote caregiver of a GTC seizure and provide a record of GTC seizure activity.
  Other Names: SPEAC System

SUMMARY:
Prospective study of an electromyography (EMG) based seizure detection and warning system for detecting generalized tonic-clonic (GTC) seizures.

DETAILED DESCRIPTION:
This study "A Pivotal, Phase III Trial of Detecting generalized tonic-clonic seizures with a Seizure Detection and Warning System in Epilepsy Patients " is a phase III, pivotal, prospective study of an electromyography (EMG) based seizure detection and warning system (tentatively named Brain Sentinel™ Seizure Detection System) for detecting generalized tonic-clonic (GTC) seizures. The detection device is worn on the bicep brachii muscles and is intended to alert a remote caregiver of a GTC seizure and provide a record of GTC seizure activity. This is to facilitate a faster intervention to the GTC seizure, and to more accurately document GTC seizure frequency in a home, skilled nursing, or inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a history of GTC seizures, either primary GTC or partial onset seizures with secondary generalization.
2. Is being admitted to a hospital for routine vEEG monitoring related to seizures.
3. Male or female between the ages of 2-99.
4. Has an upper arm circumference which is adequate for proper fit of the EMG monitor (at least 14cm).
5. If female and of childbearing potential, has a negative pregnancy test.
6. Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments.
7. Subject and/or Primary Caregiver must be competent to follow all study procedures.
8. Is able to read, speak, and understand English.

Exclusion Criteria:

1. Does not have a documented history of generalized seizures.
2. Has not had a GTC seizure within the last year AND is not expected to have a reduction of anti-epileptic drugs during their hospital admission.
3. Intracranial EEG electrodes are being used
4. The subject's upper arm circumference not adequate for proper fit of the EMG monitor (less than 14cm).
5. Pregnant female.
6. Subject/Caregiver is unable to provide consent.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and Adults with GTC seizures, either primary GTC or partial onset seizures with secondary generalization
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the Seizure Detection System | up to 1 month
  The primary outcome measure for this clinical trial will be the sensitivity of the Brain Sentinel™ Seizure Detection Systems ability to detect GTC seizure activity in comparison to a Neurologist independent review of vEEG collected in an epilepsy monitoring unit.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Szabo, MD, Principal Investigator — University Health System of San Antonio
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - University Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No